CLINICAL TRIAL: NCT02204423
Title: Upper Extremity Dysfunction Post Radial PCI: A Cohort Study Evaluating Upper Extremity Dysfunction After Percutaneous Coronary Intervention Using the Radial Artery as Access Route
Brief Title: Upper Extremity Dysfunction Post Radial Percutaneous Coronary Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albert Schweitzer Hospital (Other)
Responsible Party: Principal Investigator, Anna Koopman, MD, Albert Schweitzer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL45613.101.13
Record Dates: First submitted 2014-06-16; First posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Upper Extremity Dysfunction
Keywords: Upper extremity dysfunction; Trans-Radial Percutaneous Coronary Interventions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trans-Radial PCI (Experimental)
  Interventions: Procedure: Trans-Radial Percutaneous Coronary Intervention (TR-PCI)

INTERVENTIONS:
Procedure: Trans-Radial Percutaneous Coronary Intervention (TR-PCI)
  Other Names: Dotter-Procedure

SUMMARY:
Trans-Radial Percutaneous Coronary Intervention (TR-PCI) is rapidly becoming the gold standard. This is especially the case in primary Percutaneous Coronary Interventions (PCI), where most benefits of the radial approach, such as reduced major bleeding and mortality, can be expected. However there is very limited research available looking at the consequences of trans-radial access for upper extremity function.

The main objective of this study is to provide insight in the morbidity with regards to the upper extremity surrounding the radial access route in percutaneous coronary interventions. Secondary objectives are to provide insight in the consequences for functional status, factors influencing and financial costs of this morbidity, to identify subject who might benefit from early referral and treatment of this morbidity and to generate hypotheses for further clinical research into this matter.

The investigators hypothesis is that approximately 20% of the population will experience upper extremity dysfunction after TR-PCI.

ELIGIBILITY:
Inclusion Criteria:

* Presenting for TR-PCI at the study centre.
* The radial artery can be palpated and Doppler ultrasound examination of the radial artery shows non-occlusive flow.

Exclusion Criteria:

* Currently enrolled in another study that clinically interferes with this study and that has not passed the primary endpoint.
* The clinical condition prohibits or hinders informed consent and/or baseline examinations. E.g. cardiogenic shock and cardiopulmonary resuscitation or subconscious and semiconscious state,.
* Co-morbid condition(s) that could limit the subject's ability to participate in the study or to comply with follow-up requirements, or impact the scientific integrity of the study, e.g. loss of voluntary motor control of the studied extremities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-05 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
A binary score of upper extremity dysfunction | 2 weeks
  A positive score is defined as the presence of at least a ≥1 point increase in the Levine-Katz (Boston) questionnaire; or at least 2 of the following decreased scores compared to baseline, 2 weeks after TR-PCI:
  * ≥15% decrease in the DASH-outcome measure.
  * Increase in VAS pain score with regard to the upper extremity of ≥2 points
  * Absent signal of the radial artery using Doppler
    * 10% decrease in goniometry of the upper extremity, with a minimum decrease of 10 degree Strength
    * 60N decrease in palmar grip strength
    * 12N decrease in pinch grip strength
    * 15% decrease in isometric strength of the following manoeuvres:
      * Flexion and extension of the elbow and/or wrist
  * Sensibility loss of ≥1 filament of the hand using Semmes-Weinstein filaments according to WEST
    * 1cm increase at volumetry of the hand, using the Figure of 8-method
    * 1cm increase at volumetry of the forearm, measured circumferentially 8 cm distal of the medial epicondyle
  * Compartment syndrome

SECONDARY OUTCOMES:
Successful arterial access | During procedure
  Successful arterial access of the target radial artery, defined as the ability to successfully advance a guiding catheter and position it in the coronary ostium.
Cross-over | During procedure
  Percentage of cross-over from radial to femoral access
Anomaly | During procedure
  Presence of branching anomaly (high radial artery take-off), tortuosity (none, mild, moderate or severe), stenosis (not encountered or percentage of stenosis encountered) and/or spasm (none, mild, moderate or severe) of the radial artery
Access route complications | 6 months
  Access route complications, dissection or perforation of radial, brachial or subclavian artery, as evidenced by angiography or computed tomography
Procedural success | During procedure
  Procedural success (defined as <30% residual stenosis at the end of the procedure)
Catheter performance | During procedure
  Overall catheter performance ranging from 0 (very bad) - 5 (very good)
Procedure time | During procedure
  Procedure time in minutes, from guide catheter insertion to withdrawal
Radiation | During procedure
  Radiation time and dose, in minutes and mGy
MACCE | 6 months
  Major adverse cardiac and cerebrovascular events (MACCE), defined as:
  * Myocardial infarction (MI), according to the Third Universal definition of Myocardial Infarction
  * Target vessel revascularisation, either by PCI or surgical
  * Death
  * Cerebrovascular accident (CVA)
Bleeding | 6 months
  Bleeding events (according to Academic Research Consortium definitions) at procedure and at each consecutive follow-up
DASH | 6 months
  "Disabilities of the Arm, Shoulder and Hand" (DASH) outcome measured at two weeks, one and six months
VAS | 6 months
  Visual Analogue Scale pain score (VAS) with regard to the upper extremity at one day, two weeks, one and six months.
Occlusion | 6 months
  Presence or absence of arterial pulse when evaluating the radial artery using Doppler ultrasound examination extremity at one day, two weeks, one and six months
AROM | 6 months
  Active Range Of Motion (AROM) goniometry values in degrees of the upper extremity at two weeks, one and six months.
Strength | 6 months
  o Strength in Newton at two weeks, one and six months:
  * Palmar grip strength
  * Pinch grip strength
  * Isometric strength of the following manoeuvres:
    * Flexion and extension of the elbow
    * Flexion and extension of the wrist
Sensibility | 6 months
  Sensibility of the hand using Semmes-Weinstein filaments according to WEST at two weeks, one and six months.
Volumetry of the hand | 6 months
  Volumetry of the hand in centimeters using the Figure of eight-method extremity at one day, two weeks, one and six months.
Volumetry of the forearm | 6 months
  Volumetry of the forearm in centimetres at one day, two weeks, one and six months.
Levine-Katz (Boston) questionnaire | 6 months
  Symptom-severity score and the functional-status score of the Levine-Katz (Boston) questionnaire at two weeks, one and six months

OTHER OUTCOMES:
Hand centre | After reaching primary endpoint
  o If the primary endpoint has been reached:
  * Diagnostic procedures performed at the hand centre
  * Diagnosis of the hand centre
  * Performed treatment at the hand centre
  * Upper extremity related absence of work in days

CONTACTS AND LOCATIONS:
Locations (1):
- Albert Schweitzer Hospital, Dordrecht, South Holland, Netherlands